CLINICAL TRIAL: NCT06105619
Title: A Randomized, Controlled, Open, Multicenter, Phase II/III Clinical Study to Evaluate the Safety and Efficacy of Vebreltinib Enteric Capsules in the Treatment of sGBM/IDH Mutant Glioblastoma Patients With the ZM Fusion Gene (FUGEN).
Brief Title: A Study of PLB1001 Enteric Capsules in the Treatment of sGBM/IDH Mutant Glioblastoma Patients With the ZM Fusion Gene (FUGEN).
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beijing Pearl Biotechnology Limited Liability Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLB1001-Ⅱ-GBM-01
Record Dates: First submitted 2023-10-24; First posted 2023-10-27 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLB1001 (Experimental): Subjects will receive 300mg of PLB1001 twice daily in cycles of 4 weeks duration until death or adverse event(AE) leading to discontinuation
  Interventions: Drug: PLB1001
- Temozolomide or Cisplatin combined with etoposide (Active Comparator): Investigators can choose one of two treatments
  1. Dose density of temozolomide：100-150mg/m2/d,day 1 to 7 and day 15 to 22 of each 28-day cycle
  2. Cisplatin combined with etoposide：Cisplatin,80-100mg/m2/3 days,28 days/cycle.etoposide, 100mg/m2/d,3 days,28 days/cycle
  Interventions: Drug: Temozolomide; Drug: Cisplatin combined with Etoposide

INTERVENTIONS:
Drug: PLB1001 — PLB1001 is a capsule in the form of 300mg,twice daily.
  Other Names: Vebreltinib
  Arms: PLB1001
Drug: Temozolomide — 100-150mg/m2/d,day 1 to 7 and day 15 to 22 of each 28-day cycle
  Arms: Temozolomide or Cisplatin combined with etoposide
Drug: Cisplatin combined with Etoposide — Cisplatin:80-100mg/m2/3 days,28 days/cycle Etoposide:100mg/m2/d,3 days,28 days/cycle
  Arms: Temozolomide or Cisplatin combined with etoposide

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of PLB1001 Enteric Capsules in the treatment of PTPRZ1-MET fusion gene positive recurrent secondary glioblastoma. The main questions it aims to answer are:

1. To evaluate overall survival (OS) in the treatment of secondary glioblasts with positive recurrence of PTPRZ1-MET (ZM) fusion gene by PLB1001 Enteric Capsules.
2. To evaluate if it is safety and tolerant in the treatment of secondary glioblasts with positive recurrence of PTPRZ1-MET (ZM) fusion gene by PLB1001 Enteric Capsules.

Participants will

1. Be given PLB1001 300mg BID,oral who were randomly assigned in test group.
2. Be given Temozolomide capsules ,oral, who were randomly assigned in control group.
3. Be given EP, ivgtt, who were randomly assigned in control group.

DETAILED DESCRIPTION:
84 sGBM or IDH mutant glioblastoma patients with the ZM fusion gene will be randomly divided into group A (receive vebreltinib) or group B ( receive investigator choose), and the randomize ratio will be 1:1, patients in group A will receive PLB1001 300mg Bid, 28days/cycle. Patients in group B will receive temozolomide (100-150mg/m2/d, 7 days 1 to7 and days 15 to 22 of each 28-day cycle ) or cisplatin+etoposide(cisplatin:80-100mg/m2/3 days, 28days/cycle; etoposide:100mg/m2/d, 3days, 28 days/cycle).

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed secondary glioblastoma,or glioblastoma with IDH mutantation
2. Must have evidence of PRPRZ1-MET fusion gene positivity from the result of molecular pre-screening evaluations
3. Prior treatment with temozolomide and radiotherapy
4. Stable or decreasing dose of corticosteroids within 5 days prior to the first dose
5. Platelet count≥75×109/L,Neutrophilic granulocyte count≥1.5×109/L, Hemoglobin>90g/L,AST or ALT < 3 times the lab's upper normal limit,Serum creatinine < 1.5 times the lab's upper normal limit,INR≤2.0
6. Karnofsky performance score ≥ 60%
7. Pregnant or nursing women
8. Written consent

Exclusion Criteria:

1. Previous or current treatment with a c-Met inhibitor or HGF-targeting therapy
2. Received antibody anti-tumor drug within 30 days before enrollment
3. Previous treatment with Camustine sustained release implant
4. The subject is unable to undergo MRI scan
5. Patients with active bleeding were found by brain CT or MRI scan before enrollment
6. Uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) 150 mm Hg and/or Diastolic Blood Pressure (DBP) ≥100 mm Hg
7. Major surgery within 4 weeks prior to first dose of PLB1001
8. Pregnant or nursing women
9. Involved in other clinical trials <30 days prior to first dose

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival(OS) | 5 years
  Overall survival is defined as the time(in months)from random to the date of death.

SECONDARY OUTCOMES:
Objective Response Rate Evaluated by Investigator(ORR) | 5 years
  Objective response rate will be determined according to response assessment in neuro-oncology(RANO).
Progression Free Survival evaluated by Investigator(PFS) | 5 years
  Progression Free Survival is defined as the time (in months) from the first administration of trial treatment to the date of the first documentation of PD or death due to any cause.
Quality of Life Assessment EORTC-QLQ-C30 | 5 years
  The EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item scales and single-item measures. These include the Physical Functioning Scale and four more functional scales (role, emotional, social, and cognitive), three symptom scales (fatigue, nausea and vomiting, and pain), a global health status / QoL scale, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and difficulties). Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." The method for scoring these scales is: 1. Estimate the average of the items that contribute to the scale; this is the raw score. 2. Use a linear transformation to standardize the raw score, so that scores range from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms. A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.
Karnofsky Performance Status score | 5 years
  improved is defined as KPS increases >10 after treatment; worsen is defined as KPS decreases >10; stable is defined as KPS changes ≤10.
Quality of Life Assessment EORTC-QLQ-BN20 | 5 years
  The EORTC-QLQ-BN20 covers future uncertainty, visual disorder, motor dysfunction, communication deficit, headache, seizures, drowsiness, hair loss, itching, difficulty with bladder control, and weakness of both legs. Patients respond by self-report, with most items rated on a 4-point scale, from 1 "not at all" to 4 "very much", except for the two global health status/quality of life items, which are measured on a 7-point Likert scale ("very poor" through "excellent"). The method for scoring these scales is: 1. Estimate the average of the items that contribute to the scale; this is the raw score. 2. Use a linear transformation to standardize the raw score, so that scores range from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms. A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Li, Principal Investigator — Beijing Tiantan Hospital; Xiaoguang Qiu, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No